CLINICAL TRIAL: NCT05267288
Title: Phase II Study of Afatinib Plus Bevacizumab in the Treatment Epidermal Growth Factor Receptor (EGFR) Exon G719X, S768I, and L861Q Mutation Metastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QDCH2022-02-18
Record Dates: First submitted 2022-02-17; First posted 2022-03-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: PFS
MeSH Terms: interventions — Afatinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- afatinib plus bevacizumab (Experimental): afatinib 40mg oral continually bevacizumab 15mg/kg, iv day 1, every 21days until disease progression, untolerated toxicities of patient death.
  Interventions: Drug: afatinib

INTERVENTIONS:
Drug: afatinib — afatinib 40mg oral, bevacizumab 15mg/kg iv, every 21days, until progression disease, untolerated toxicities, or patient death.
  Other Names: bevacizumab

SUMMARY:
There is no report afatinib plus bevacizumab in the treatment of EGFR G719X, S768I, and L861Q single or compond mutation of metastatic non-small-cell lung cancer (NSCLC). The purpose of this study is to study afatinib combined with bevacizumab in the management of it.

DETAILED DESCRIPTION:
Lung cancer is one of the most common types of cancer and is the most common cause of death from cancer (almost 20 percent [%] of cancer deaths); NSCLC accounts for 80% to 85% of lung cancers. The hypothesis is that afatinib plus bevacizumab in patients with metastatic NSCLC characterized by EGFRuncommon mutations with G719X, S768I, and L861Q. Efficacy assessments will include disease assessment, symptomatic progression and patient-reported outcome. Safety assessments will include physical examinations, vital signs, electrocardiograms (ECGs), Eastern Cooperative Oncology Group (ECOG) performance status and clinical safety laboratory assessments (serum chemistry, hematology, coagulation, and urinalysis).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed, locally advanced or metastatic, nonsquamous non-small cell lung cancer (NSCLC) with documented primary epidermal growth factor receptor (EGFR) Exon G719X, S768I, L861Q mutation Participant must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Participant must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, or 2 Participant must agree to genetic characterization of tumor status through the required pretreatment tumor biopsy (or submission of equivalent archival material), as well as baseline and periodic blood samples for analysis of tumor mutations in the bloodstream A female participant of childbearing potential must have a negative serum or urine test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study

Exclusion Criteria:

Participant has history of spinal cord compression that has not been treated definitively with surgery or radiation Participant has a medical history of interstitial lung disease (ILD), including drug-induced ILD, or radiation pneumonitis Participant has a contraindication to the use afatinib or Bevacizumab

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | up to 18 months
  Progression-Free Survival (PFS) According to RECIST v1.1 as Assessed by Blinded Independent Central Review (BICR)

SECONDARY OUTCOMES:
overall survival | Up to 48 months ]
  Overall Survival is defined as the time from the date of randomization to the date of participant's death due to any cause.
Objective Response Rate (ORR) | up to 18 months
  ORR is defined as the percentage of participants who achieve either a complete response (CR) or partial response (PR) as defined by BICR using RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Qingdao Central Hospital, Qingdao, Shandong
  - Qingdao Central Hospital, Qingdao

IPD SHARING:
Plan to Share IPD: No